CLINICAL TRIAL: NCT07000825
Title: EFFECTS OF INGESTING AN EXTRACT OR YERBA MATE (ILEX PARAGUARIENSIS) ON NUTRICIONAL, METABOLIC AND INFLAMMATORY PARAMETERS AND OXIDATIVE STATUS IN OVERWEIGHT INDIVIDUALS
Brief Title: EFFECTS OF A YERBA MATE EXTRACT IN REDUCING METABOLIC SYNDROME IN OVERWEIGHT INDIVIDUALS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal da Fronteira Sul (Other)
Collaborators: Itaipu Technological Park (ITP) (Network); Fundação Araucária (Other)
Responsible Party: Principal Investigator, Eloá Angélica Koehnlein, Professor, Universidade Federal da Fronteira Sul
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 84742724.6.0000.5564
Record Dates: First submitted 2025-03-17; First posted 2025-06-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Metabolic Syndrome; Diabetes; Oxidative Stress; Dyslipidemia; Inflamation
Keywords: glycemic control; lipid metabolism; oxidative stress; metabolic syndrome; adipose tissue
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Dyslipidemias | interventions — Methods

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, parallel-group clinical trial with a 90-day intervention. The trial will be registered with the Brazilian Clinical Trial Registry - Ministry of Health (https://ensaiosclinicos.gov.br/) and will be conducted in accordance with the CONSORT guidelines (Schulz KF, Altman DG, Moher D, for CONSORT Group. CONSORT Statement 2010: updated guidelines for reporting parallel-group randomized trials). The clinical trial will be conducted from March 2025 to July 2026.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (yerba mate) (Experimental): 2,250 mg of standardized yerba mate extract will be administered in 9 capsules, 3 times a day, just before the main meals.
  Interventions: Dietary Supplement: Intervention with yerba mate extract or placebo
- Test (yerba mate) (Placebo Comparator): 9 capsules containing maltodextrin will be administered 3 times a day, just before the main meals.
  Interventions: Dietary Supplement: Intervention with yerba mate extract or placebo

INTERVENTIONS:
Dietary Supplement: Intervention with yerba mate extract or placebo — The standardized extract of yerba mate (Ilex paraguariensis) will be supplied by Sustentec. It is a dry extract of the plant's green, powdered leaves, obtained through aqueous extraction. The extract was obtained by infusing the dried leaves of the plant and the drying process was carried out using a spray-dryer (ratio 6/1 leaves/extract). The extract will be encapsulated containing 250 mg each. Administration Intervention group: 2,250 mg of standardized yerba mate extract will be administered in 9 capsules, 3 times a day, just before the main meals. This amount will provide approximately 980 mg of caffeoylquinic acids/day, which was defined based on the estimated usual intake of caffeoylquinic acids by individuals in a municipality in the southern region of the country, from traditional drinks made with yerba mate (chimarrão and tereré) (Gebara et al., 2017). Placebo group: 9 capsules containing maltodextrin will be administered 3 times a day, just before the main meals.

SUMMARY:
Yerba mate (Ilex paraguariensis), a traditional drink consumed in different parts of the word, but especially in southern Brazil, is an importante source of polyphenols and has a high antioxidant potencial, With a moderate content of methylxanthines, yerba mate has stood out for its promising effects in modulating metabolic pathways in pre-clinical models. However, its beneficial effets in clinical trials have yet to be elucidated. Overweight and chronic non-communicable diases are urgent public health conditions and reducing the risk of these conditions through food sources is one of the most sustainable approaches. This study aims to evaluate the impact of a standardized extract of yerba mate on nutritional, biochemical, metabolic, inflammatory and antioxidant status parameters in overweight individuals compared to a placebo. A double-blind, parallel, randomized, placebo- controlled clinical trial will be conducted involving 80 overweight individuals. The subjects will receive an encapsulated yerba mate extract totaling 2,250 mg or a corresponding placebo, fractionated three times a day. This amount was defined according to previous studies thet estimated the habitual intake of yerba mate in the form of chimarrão or tererê by adults in a city in the southern region of the country. Anthropometric measurements, composition, blood pressure and blod and stool samples will be collected for nutritional assessment, metabolic and inflammatory parameters and antioxidant status assessment on days 0 and 90. The data will be analyzed descriptively and inferentially. Differences in the individuals characteristics at baseline and comparisons between groups will be aseessed using the difference of means test (depending on the normality of the data) and chi-square or Fisher-s exact test for categorical variabes, In addition, to compare the effect of the intervention between the groups, a two-way analysis of covariance will be used. A 5% significance level will be adopted. It is expect to find positive effects of yerba mate extract on the parameters assessed.

ELIGIBILITY:
Inclusion Criteria:

1. men and women;
2. aged between 40 and 65 years;
3. with no previous cardiovascular history;
4. individuals who are non-smokers or who have stopped smoking in the last 3 years;
5. individuals who agree to maintain a habitual diet and physical activity;
6. individuals who agree to maintain habitual consumption of polyphenol-rich beverages (yerba mate, teas, coffee, wine, cocoa, soy milk and fruit juice) during the course of the study;
7. individuals who are not taking hypoglycemic, antihypertensive or anticholesterolemic drugs and;
8. individuals who are overweight or obese (BMI≥25 to 34 Kg/m2 );
9. individuals who have given up nutritional monitoring at least 3 months or who are undergoing nutritional treatment, but who are not showing weight changes of >5% in the last 3 months.

Exclusion Criteria:

1. diagnosis uncontrolled metabolic or endocrine pathologies;
2. who have undergone obesity surgery;
3. post-menopausal women;
4. pregnant and breastfeeding women;
5. use of antipsychotics;
6. with a vegetarian or vegan diet;
7. who use probiotics and food supplements with antioxidant characteristics;
8. those who have had a weight change of more than 10% in the last 3 months; 9) in treatment for excess body weight (hypocaloric diet or current nutritional treatment);

10) smokers or chronic alcoholics; 11) Severe hypertension, history of cardiovascular disease with clinical complications such as: acute myocardial infarction and other coronary heart disease; 12) individuals with known malignant neoplasms, gastrointestinal diseases, kidney disease and/or liver disease.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
body mass index | 12 weeks
  measured by weight in kilograms and height in meters
fat percentage | 12 weeks
  measured by electrical bioimpedance
diabetes | 12 weeks
  measured by plasma glucose
abdominal fat | 12 weeks
  measured by waist circumference
dyslipidemia | 12 weeks
  measured by lipid profile
diabetes | 12 weeks
  measured by insulin levels

SECONDARY OUTCOMES:
inflamation | 12 weeks
  measured by cytokine levels
oxidative stress | 12 weeks
  measured by lipid peroxidation
oxidative stress | 12 weeks
  measured by plasma thio levels
oxidative stress | 12 weeks
  measured by total antioxidant capacity of plasma
transcriptome | 12 weeks
  measured by gene expression
gut microbiota | 12 weeks
  measured by microbiome DNA

CONTACTS AND LOCATIONS:
Overall Officials: Eloá A Koehnlein, Doctorate, Principal Investigator — Universidade Federal da Fronteira Sul
Locations (1):
- Universidade Federal da Fronteira Sul, Realeza, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No